CLINICAL TRIAL: NCT02441452
Title: Functional Capacity of Exercise and Lung Function in Patients Submitted to Early Rehabilitation Program After Nuss Procedure: a Randomized Controlled Trial
Brief Title: Functional Capacity of Exercise and Lung Function in Patients Submitted Early Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Coracao (Other Government)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Sâmia Geórgia Dantas Linhares, Physiotherapist, Instituto do Coracao
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: InCor Heart Institute
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Funnel Chest
Keywords: Nuss procedure; postoperative care; early ambulation
MeSH Terms: conditions — Funnel Chest | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early rehabilitation (Active Comparator): one day before surgery, patients and their families were instructed by physiotherapists than explained the importance to perform physical exercises and breath exercises in postoperative. At the postoperative recovery room, after extubation and fully awake, patients started physiotherapy exercises, as physical exercises of moving up upper and lower extremities accompanied by deep breathing exercises. After than, the patients standed up beside the bed and if there was no complications, patients performed ambulation.
  Interventions: Other: Early rehabilitation
- Conventional care (No Intervention): Usual care routine postoperative.

INTERVENTIONS:
Other: Early rehabilitation — The physical exercises and breathing exercises are started as soon as after the Nuss procedure
  Other Names: Physical exercises and breathing exercises after surgery
  Arms: Early rehabilitation

SUMMARY:
The aim of this study was to compare the functional capacity of exercise by six-minute walk test and lung function by spirometry, before and after Nuss procedure in subjects who have undergone the early rehabiliation program with those who were under conventional care. Researchers want to find out if early rehabilitation is a strategy to enhance recovery after Nuss procedure.

DETAILED DESCRIPTION:
The replacement of some traditional approaches in surgical care has demonstrated that surgical recovery can be accelerated and convalescence decreased. These multimodal approaches focuses on enhancing recovery and reducing morbidity by reduction of surgical stress,minimal invasive surgery, optimized pain relief, early nutrition and ambulation.

In postoperative, the bed rest leads to the increase in muscle loss and weakness, impairs pulmonary function, predisposes to venous stasis and thromboembolism, increases infection complications and reduces functional capacity even in patients who are not restricted to bed.

However, few studies have focused on when start the mobilization and which effects on functional capacity of exercise and lung function during hospital stay.

In this trial the investigators will consider early rehabilitation to be safe and feasible in Nuss procedure.

ELIGIBILITY:
Inclusion Criteria:

* children who are scheduled to undergo a surgical procedure for the correction of pectus excavatum
* sign the informed consent form
* independent ambulation
* ability to understand and follow instructions
* ability to perform lung function test

Exclusion Criteria:

* contraindications for epidural catheter placement
* patients undergoing the open surgical repair of pectus excavatum
* refusal to do physical exercises on postoperative
* patients did not perform the six-minute walk test and lung function test on postoperative

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Functional capacity of exercise ( six-minute walk test) | participants will be followed for the duration of hospital stay, an expected average of 6 days
  Change from baseline in distance walking on hospital discharge
Lung function (spirometry) | participants will be followed for the duration of hospital stay, an expected average of 6 days
  Change from baseline in lung function on hospital discharge

SECONDARY OUTCOMES:
Time to first postoperative ambulation | up 2 hour after surgery
  Time from end of surgical procedure until first postoperative ambulation was used as an indicator for early rehabilitation.
Pain intensity | participants will be followed for the duration of hospital stay, an expected average of 6 days
  Auto-evaluation of pain (the numeric rating scale and visual analogue scale of pain from 0 -no pain- to 10 - maximal pain)
The length of hospital stay | expected average of 6 days
  Time to achieve standardized hospital discharge criteria (tolerance of oral intake, recovery of lower gastrointestinal function, adequate pain control on oral analgesia, ability to mobilize and self care and no evidence of complications or untreated medical problems).